CLINICAL TRIAL: NCT03904797
Title: Colorado Early Intervention Outcomes Research Using Innovative Patient-Reported Outcome (PRO) Measures
Brief Title: Electronic Patient-reported Outcomes (e-PROs) in Early Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Rocky Mountain Human Services (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-0139
Record Dates: First submitted 2019-03-25; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-03

CONDITIONS: Developmental Disability; Development Delay
Keywords: patient-reported outcome; electronic; participation; early intervention
MeSH Terms: conditions — Developmental Disabilities; Learning Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- e-PRO (Experimental): EI service coordinators participated in a 90-minute training on the study protocol, to gain clearance to recruit families when they were being contacted to schedule their annual reviews of progress. The recruitment protocol was later modified in response to low enrollment, such that a designated EI staff member was paired with research staff to recruit participants. Eligible and interested caregivers visited the project website to create an account, confirmed study eligibility, provided informed consent and HIPAA authorization for abstracting select EI service use data, and completed a demographic questionnaire and the Young Children's Participation and Environment Measure (YC-PEM) e-PRO. Caregivers received immediate access to an online report summarizing their e-PRO responses to share with their child's EI team
  Interventions: Behavioral: Young Children's Participation and Environment Measure (YC-PEM) electronic patient-reported outcome (e-PRO)

INTERVENTIONS:
Behavioral: Young Children's Participation and Environment Measure (YC-PEM) electronic patient-reported outcome (e-PRO) — Participants were primary caregivers (n=149) recruited from a large, urban early intervention program. All caregivers were approached by early intervention staff the month prior to the child's annual evaluation of progress.
  Each caregiver confirmed his or her eligibility online by verifying that they were at least 18 years old; could read, write, and speak English or Spanish; had internet access; and had a child between 0-3 years old who had received early intervention for at least 3 months.
  Participants enrolled online and provided consent, signed a HIPAA authorization for service record release, and then proceeded to completing a demographic questionnaire and YC-PEM e-PRO to receive an online report of their responses to share with their child's EI team.

SUMMARY:
A major goal of early intervention (EI) is to employ a family-centered approach to helping children to optimally function at home and in the community. However, the effects of EI are poorly understood. The aims of this project are: 1) to test the feasibility, acceptability, and value of introducing novel electronic patient-reported outcome (e-PRO) measures in EI, to strengthen family-centered EI care; and 2) to obtain and pair these outcomes data with EI program data, to further determine the value of e-PRO data collection for examining links between EI service use and functional outcomes among families who are enrolled in a large, urban EI program.

DETAILED DESCRIPTION:
Approximately 5,800 infants and toddlers with developmental disabilities (e.g., cerebral palsy, Down syndrome, complex chronic conditions) and delays access Early Intervention Colorado (EI-CO) annually. A primary goal of EI-CO is to employ a family-centered care approach to help children optimally function at home and in the community. Hence, early intervention is a common source of rehabilitation (i.e., physical, occupational, speech and language therapy) for EI-CO eligible families.

However, the effects of EI-CO are poorly understood. Numerous challenges exist with obtaining EI-CO outcomes data, including a paucity of validated and feasible functional outcome measures for use in EI outcomes reporting. These challenges have resulted in inadequate knowledge about EI service use and outcomes to guide service delivery. Despite these challenges, recent policy changes have resulted in EI-CO service providers being pressed to ensure high quality care with limited resources and evidence to guide their clinical decision-making about effective and efficient interventions. This proposal addresses the need to fill critical knowledge gaps about the adequacy of EI services with an eye toward improving care quality.

This study involves families who have/are receiving EI-CO services through Rocky Mountain Human Services (RMHS), the largest EI program in Denver Metro. The purpose of this study is to test the feasibility, acceptability, and value of collecting electronic patient-reported outcomes (e-PRO) data to engage families when their child is due for an annual evaluation of progress. To further demonstrate the value of e-PRO data collection, these data will be paired with program data to estimate the association between EI-CO service use and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver is at least 18 years old;
* Caregiver can read, write, and speak English or Spanish;
* Caregiver had internet access;
* Caregiver has a child between 0-3 years old who had received early intervention at RMHS for at least 3 months.

Exclusion Criteria:

* Caregiver is less than 18 years old
* Caregiver reads, speaks, and writes in a language other than English or Spanish
* Caregiver does not have internet access
* Caregiver has a child who has received EI services for less than 3 months
* Caregiver has a child older than 3 years (36 months)

Ages: 1 Month to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 149 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
YC-PEM e-PRO Feasibility as assessed by enrollment rate | up to 4 weeks
  Enrollment rate was estimated as the proportion of eligible participants who enrolled in the study. The success of feasibility was determined as e-PRO enrollment rates of 50% or higher based on what is known about the percentage of families who opt into family assessment as part of usual care.
YC-PEM e-PRO Acceptability as assessed by caregiver perceptions of overall helpfulness | up to 4 weeks
  Caregiver responses to an open-ended item were coded into a one of three categories (yes, helpful; somewhat helpful; not helpful) to create a new variable that captured the extent to which caregivers perceived the YC-PEM e-PRO to be useful for planning EI care.
YC-PEM e-PRO Value as assessed by proportion of participants viewing e-PRO online report | up to 4 weeks
  The percentage of participants who viewed a summary of their e-PRO responses via an online report was estimated.
YC-PEM e-PRO Feasibility as assessed by completion rate | up to 4 weeks
  Feasibility was determined as the proportion of participants who enrolled that completed the YC-PEM e-PRO. The success of feasibility was determined as completion rates of 50% or higher based on family assessment completion rates within usual care.
YC-PEM e-PRO Feasibility as assessed by completion time in minutes and seconds | up to 4 weeks
  The success of feasibility was determined as e-PRO completion time of less than 45 minutes based on family assessment completion time within usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Mary A Khetani, ScD, Principal Investigator — Board of Trustees at University of Illinois

IPD SHARING:
Plan to Share IPD: Yes
NIH funds were secured to archive a subset of the data as a restricted use data file, and the dataset is being curated now.
Supporting Information: Study Protocol
Time Frame: The subset of data are expected to become publicly available as of June 2019, but it not yet known for how long the data will be available.
Access Criteria: The criteria for access is being developed at this time and will be updated when finalized.

REFERENCES:
- [Derived] Albrecht EC, Kaelin VC, Rigau BL, Dooling-Litfin JK, Scully EA, Murphy NJ, McManus BM, Khetani MA; High Value Early Intervention Research Group. Pilot implementation of an electronic patient-reported outcome measure for planning and monitoring participation-focused care in early intervention. BMC Med Inform Decis Mak. 2020 Aug 24;20(1):199. doi: 10.1186/s12911-020-01189-9. PMID 32838772
- [Derived] Khetani MA, McManus BM, Albrecht EC, Kaelin VC, Dooling-Litfin JK, Scully EA; High Value Early Intervention Research Group. Early intervention service intensity and young children's home participation. BMC Pediatr. 2020 Jul 3;20(1):330. doi: 10.1186/s12887-020-02182-x. PMID 32620161